CLINICAL TRIAL: NCT02469779
Title: Middle and High School Students' Reactions to a Health Interactive Website: ASPIRE Reactions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-0296
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Tobacco Use Cessation; Tobacco Prevention
Keywords: Tobacco Prevention; ASPIRE Website; Surveys; Questionnaires; Focus Groups; Health Interactive Website
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASPIRE Group (Experimental): Participants complete baseline survey. Participants view the ASPIRE website containing videos, activities, and health information facts about the effects of smoking, the benefits of meditation, and healthy living. This viewing will be videotaped and audio recorded. 3 to 4 sessions will be completed. After each website session, survey will be completed.
  Interventions: Behavioral: Surveys; Behavioral: ASPIRE Website; Behavioral: Follow Up Survey
- Control Group (Active Comparator): Participants complete baseline survey. Participants view the ASPIRE text-based website containing health information facts about smoking, the benefits of meditation, and healthy living. This viewing will be videotaped and audio recorded. 3 to 4 sessions will be completed. After each website session, survey will be completed.
  Interventions: Behavioral: Surveys; Behavioral: ASPIRE Text-Based Website; Behavioral: Follow Up Survey

INTERVENTIONS:
Behavioral: Surveys — At baseline participants complete survey about their mental and physical health and their opinions concerning health information and the internet. The survey will take about 15-20 minutes to complete.
  Other Names: Questionnaires
Behavioral: ASPIRE Website — Participants view the ASPIRE website containing videos, activities, and health information facts about the effects of smoking, the benefits of meditation, and healthy living. This viewing will be videotaped
  Arms: ASPIRE Group
Behavioral: ASPIRE Text-Based Website — Participants view the ASPIRE text-based website containing health information facts about smoking, the benefits of meditation, and healthy living.
  Arms: Control Group
Behavioral: Follow Up Survey — Participants complete a follow-up survey about their opinions concerning health information and the internet immediately after they have completed their last session on the website.
  Other Names: Questionnaire

SUMMARY:
The goal of this research study is to learn how middle and high school students react to an interactive website called ASPIRE ( A Smoking Prevention Interactive Experience) and health information online and what their preferences are when using ASPIRE.

Researchers hope to use the results of this study to design more effective online health programs to provide middle and high school students with up-to-date information about tobacco use, meditation, and general health and well-being.

DETAILED DESCRIPTION:
Participants complete up to 2 separate parts.

Part 1:

For Part 1, participants complete a survey about their mental and physical health and their opinions concerning health information and the internet. The survey takes about 15-20 minutes to complete.

Part 2:

If the results of the survey show eligibility, participants complete Part 2 of the study. For Part 2 participants are randomly assigned (as in a roll of dice) to 1 of 2 study groups. Participants have a 1 in 3 chance of being assigned to receive standard care. Participants have a 2 in 3 chance of being assigned to use the ASPIRE website. This is done because no one knows if one study group is better, the same, or worse than the other group.

If participant assigned to receive standard care, he or she is shown a website that has the same information presented in ASPIRE, but in text form.

Participants in both groups sit in front of a computer and go onto a website. Both the ASPIRE website and the text-based website have been designed for middle and high school students. The ASPIRE website has videos, activities, and health information facts about the effects of smoking, the benefits of meditation, and healthy living. The text-based website only has health information facts about smoking, the benefits of meditation, and healthy living. Participants complete 3 to 4 sessions using either the ASPIRE website or the text-based website throughout their first semester. Each session lasts about 40 minutes.

The use of the websites will be videotaped.

Follow-Up Surveys:

Participants complete a follow-up survey about their opinions concerning health information and the internet immediately after they complete their last session on the website. The follow-up surveys take about 15 minutes to complete.

Length of Study:

Active participation on this study is over after participants complete the follow-up survey. If participant does not continue onto Part 2 of the study, their active participation is over after they complete Part 1 of the study.

Other Information:

Participants take part in this study at their school during their after school program.

During the use of the website, each study participant is individually videotaped and audio recorded. The videotapes and audio recordings are used to help the research staff analyze each participant's use of the websites. The video tapes and audio recordings are stored on a password-protected encrypted hard drive that is stored in a locked office at MD Anderson. Only the study researcher and authorized members of the research staff are allowed to use the videotapes and audio recordings (for research purposes).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 11 through 18 (11 and 18 included)
2. High school and Middle School students are both eligible
3. All 150 are nonsmokers. Nonsmokers are defined as individuals who have not smoked, not even part of a cigarette in the past year.
4. All will score above the median on smoking susceptibility
5. 10 will be White/Caucasian participants, 5 will be African American participants, 10 will be Hispanic participants, and 5 will be Asian participants.
6. English speaking

Exclusion Criteria:

1)None

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 700 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Intention to Smoke | 1 day
  This outcome is measured using the validated susceptibility to smoke scale in a Likert scale format and baseline and immediate follow up.

SECONDARY OUTCOMES:
Emotional Response | 4 days
  Outcome measured using validated Likert scales. In addition, facial expressions of happiness, sadness, disgust, fear, anger, and surprise are measured using a software program of emotion recognition for facial movement. The software captures the extent of expression of each of the emotions on a scale from 0 to 1.
Participants' Reported Qualitatively Attributes in ASPIRE | 1 day
  Participants' reported qualitatively attributes (i.e. features) in ASPIRE that they recall to be emotionally involving. This report conducted using open-ended questions.
Relationship Between Emotional Involvement During Use of ASPIRE Website and Change in Susceptibility to Smoking | 1 day
  Generation of emotional expression during use of ASPIRE is dependent on data for use of ASPIRE features, and data for emotional expression. Recorded videos of participant's online behavior analyzed via manual content analysis. Recorded videos of online behavior (i.e. mouse movement on the screen, clicking, dragging behaviors, and what the webpage presents) also analyzed using N-vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Prokhorov, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Mt. Calvary Baptist Church, Houston, Texas
  - Young Men's Christian Association (YMCA), Houston, Texas

REFERENCES:
- [Derived] Khalil GE, Wang H, Calabro KS, Mitra N, Shegog R, Prokhorov AV. From the Experience of Interactivity and Entertainment to Lower Intention to Smoke: A Randomized Controlled Trial and Path Analysis of a Web-Based Smoking Prevention Program for Adolescents. J Med Internet Res. 2017 Feb 16;19(2):e44. doi: 10.2196/jmir.7174. PMID 28209560
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org